CLINICAL TRIAL: NCT05930379
Title: A Feasibility Pilot Study on Lee Silverman Voice Treatment (LSVT)-Loud on Voice Intensity and Voice Use in Daily Living in People With Multiple Sclerosis: a Telerehabilitation Approach
Brief Title: A Feasibility Pilot Study on Lee Silverman Voice Treatment-Loud: a Telerehabilitation Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ON-LOUD
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Telerehabilitation; Speech Therapy; Multiple Sclerosis; Voice Intensity; Hypophonia; Digital Health
MeSH Terms: conditions — Multiple Sclerosis; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSVT-Loud delivered by telerehabilitation (Experimental): F - Frequency: 7 times/week for 4 weeks according to a mixed model (4 days of synchronous sessions followed by independent practice + 3 asynchronous sessions); I - Intensity: sessions customized according to the patient's functional abilities to ensure the progression of difficulty in rehabilitation sessions; T- Time: each synchronous session will last about 60 minutes, each independent practice will last about 5-10 minutes, and each asynchronous session will last about 30 minutes; T- Type: Individual speech therapy sessions with the Lee Silverman Voice Treatment-Loud method delivered by telerehabilitation.
  Interventions: Other: LSVT-Loud delivered by telerehabilitation
- LSVT-Loud in the clinic (Active Comparator): The frequency, intensity, time of the rehabilitation sessions will be the same as the experimental group.
  T- Type: Individual speech therapy sessions with the Lee Silverman Voice Treatment-Loud method delivered in the clinic.
  Interventions: Other: LSVT-Loud in the clinic

INTERVENTIONS:
Other: LSVT-Loud delivered by telerehabilitation — LSVT-Loud treatment delivered by telerehabilitation
  Arms: LSVT-Loud delivered by telerehabilitation
Other: LSVT-Loud in the clinic — LSVT-Loud delivered face-to-face in the clinic
  Arms: LSVT-Loud in the clinic

SUMMARY:
Multiple Sclerosis (MS) is one of the most common causes of neurological disability in young adults. At least 62% of people with MS have speech, vocal, or communication disorders. Among these, alterations in voice intensity and quality constitute a limitation in MS people's social life leading to experience difficulties in work, conversations, and communication especially in noisy environments or through the telephone. Though voice and speech impairments and speech impairments are widely prevalent in this population, only 2% of the people receive speech therapy. The Lee Silverman Voice Treatment (LSVT)-Loud is a well-documented, efficacious intensive speech intervention, for treating hypophonia in subjects with neurological conditions. Despite the effectiveness of LSVT-Loud treatment on the voice has been reported in MS, several factors prevent the agile use of this method in rehabilitation centers: motor disability, work commitments, and distance barriers may preclude repeated attendance of this intervention at a healthcare facility. Telerehabilitation represents a feasible solution to bypass these potential barriers related to attendance at the rehabilitation programs in the clinic. The increasing evidence sustains the role of telerehabilitation for the migration of care from the clinic to the patient's homes, overcoming several obstacles affecting service accessibility. Previous studies showed the validity and the non-inferiority of LSVT-Loud delivered via telerehabilitation in subjects with Parkinson's Disease, while no pieces of evidence are still available on the efficacy of voice treatment delivered by telerehabilitation in MS. It is plausible to assume that LSVT-Loud delivered by telerehabilitation would be feasible and provide a beneficial effect also for MS non-inferior compared to the same treatment delivered in the clinic.

DETAILED DESCRIPTION:
20 patients with MS will be recruited from IRCCS Fondazione Don Carlo Gnocchi ONLUS, Milan, according to inclusion/exclusion criteria detailed in the "Eligibility Criteria" section.

Participants will be randomized into 2 different groups:

Group 1: Lee Silverman Voice Treatment - Loud delivered by telerehabilitation at home (Experimental group); Group 2: Lee Silverman Voice Treatment - Loud delivered in the clinic (Control group).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS according to the criteria of MC Donald 2010 (Polman et al., 2011; Thompson et al., 2018)
* perceived voice intensity disability and severity of speech and voice disorder prior to treatment (as judged independently by two speech-language pathologists highly experienced with voice and motor speech disorders)
* age ≥ 18;
* not treated for hypophonia in the six months before enrollment in the study
* with a preserved cognitive level at the Mini-Mental State Examination (MMSE test >24) (Folstein et al., 1975);
* available and able to use a PC with an internet connection at home to access the telerehabilitation sessions;
* agreeing to participate with the signature of the informed consent form;
* stable drug treatment (last 3 months), if any;
* absence of relapses (last month) before taking part in the study.

Exclusion Criteria:

* presence of dysphonia related to other diseases;
* presence of other neurological disorders different from MS;
* presence of major psychiatric conditions;
* presence of severe impairment of visual and/or acoustic perception;
* history of laryngeal cancer, radiotherapy, or head-neck trauma, or intubation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in the vocal Intensity during 1-minute monologue dB SPL | Baseline, post-treatment (up to 4 weeks)
  Participants will be requested to speak about daily activities at a comfortable frequency and intensity level. A specific task identical for each participant will be given: "Please speak for at least a minute." For monologue (and other acoustic variables described below) recording setup follows published recommendations, mouth-to-microphone distance is kept at 30 cm and we will calculate the mean of the first three recordings and PRAAT software (www.praat.org) will be used to record and analyze voice parameters.

SECONDARY OUTCOMES:
Change in the vocal Intensity during 1-minute monologue dB SPL | follow-up (up to 6 months from the end of the treatment)
  Participants will be requested to speak about daily activities at a comfortable frequency and intensity level. A specific task identical for each participant will be given: "Please speak for at least a minute." For monologue (and other acoustic variables described below) recording setup follows published recommendations, mouth-to-microphone distance is kept at 30 cm and we will calculate the mean of the first three recordings and PRAAT software (www.praat.org) will be used to record and analyze voice parameters.
Change in sustained /a/ voice intensity (dB SPL/a/) | Baseline, post-treatment (up to 4 weeks) and follow-up (up to 6 months from the end of treatment)
  Participants' voices will be monitored for a total of 4 hours of consecutive speech. Voice data from daily life will be registered using the Vocal Holter Med (VHM) before and after the interventions. VHM consists of a contact microphone placed in a collar worn around the neck as well as a device for data storage that can be worn in a pocket during the day. The contact microphone measures the skin vibrations caused by the activity of the vocal cords. Besides the voice indicators, also local temperature and relative humidity are measured during monitoring.
Change in the perception of voice as measured by the Voice Handicap Index (VHI, Jacobson et al., 1997) | Baseline, post-treatment (up to 4 weeks) and follow-up (up to 6 months from the end of treatment
  VHI is a standardized 30-point questionnaire, divided into three subscales covering functional, emotional, and physical aspects of voice disorders. Participants have to rate each statement using a 5-point scale scored from 0 (never) to 4 (always); the maximum score is 120 (worst score). The value of 12 points on the VHI test should be considered as a threshold for rating the handicap caused by voice disorders.
hange in perceived quality of life (especially in cognition, life activities, and participation domain) as measured by the World Health Organization disability assessment schedule 2.0 (WHODAS 2.0; Federici et al., 2017) | Baseline, post-treatment (up to 4 weeks) and follow-up (up to 6 months from the end of treatment
  WHODAS 2.0 covers six domains of functioning including Cognition, Mobility, Self-care, Getting along, Life activities, Participation. Scores assigned to each item are on a 5-point scale ranging from (0) "none" to (4) "extreme" with higher scores indicating a higher disability. The 36-item version will be administered and both summary scores (score range 0-144 with higher numbers indicating higher disability) and domain-specific scores for the six different functioning domains (especially in cognition, life activities, and participation domain; score range 0-24 for each domain with higher numbers indicating higher disability) will be considered.
Protocol adherence | post-treatment (up to 4 weeks)
  Synchronous sessions' adherence to the treatment will be registered by the telerehabilitation platform (experimental group) or by the therapist (control group). Asynchronous sessions' attendance will be registered by the completion of the patient's diary.

OTHER OUTCOMES:
Technological Systems interaction perceived experience as measured by the User Experience Questionnaire (UEQ; Schrepp et al., 2017) | post-treatment (up to 4 weeks)
  The UEQ is a 26-item scale (semantic differential scale: each item consists of two opposite adjectives, e.g., boring vs. exciting) that allows calculating six different domains: (1) attractiveness (overall impression of the system), (2) perspicuity: easily to learn how to use the system; (3) efficiency (user's effort to solve tasks); (4) dependability (feeling of control of the interaction); (5) stimulation (motivation to use the system); and (6) novelty (innovation and creation of system). The mean of the item score of each domain will be standardized based on a data benchmark (Schrepp et al., 2017).
Intrinsic Motivation in the rehabilitation program as measured by the Intrinsic Motivation Inventory - Interest/Enjoyment subscale (IMI-IE; McAuley et al., 1989) | post-treatment (up to 4 weeks)
  IMI-IE consisted of a pool of 7 items with a 7 points Likert scale ranging from (1) "Absolutely Not" to (7) "Absolutely Yes". A total score (average of the item scores) will be considered.
Number of adverse events | post-treatment (up to 4 weeks)
  Adverse events will be listed in the patient's diary considering both events occurring during the therapy and those occurring outside of the sessions but within the rehabilitation protocol period
4. Perceived rehabilitation engagement, acceptability, feasibility, frequency, and dose adequacy | post-treatment (up to 4 weeks)
  Individual and group ad-hoc interviews will be performed during and after the rehabilitation protocol period.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Gnocchi ONLUS, Milan, Italy/Milan, Italy